CLINICAL TRIAL: NCT04996446
Title: Safety and Efficacy of the Combinationg of Associating Liver Partition and Portal Vein Ligation for Staged Hepatectomy (ALPPS) and Tislelizumab in Liver Malignancy
Brief Title: ALPPS Combined With Tislelizumab in Liver Malignancy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Head of liver surgery department, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-183-2103
Record Dates: First submitted 2021-08-04; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Liver Malignant Tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alpps plus Tislelizumab group (Experimental): Patients who meet the inclusion criteria will receive ALPPS stage I surgery, treated with Tislelizumab 2-4 weeks after stage I surgery, and receive ALPPS stage II surgery 2-4 weeks after Tislelizumab treatment, and treated with Tislelizumab q3W 6-12 months after stage II surgery.
  Interventions: Drug: Tislelizumab; Procedure: ALPPS surgery
- Alpps group (Active Comparator): Patients who meet the inclusion criteria will receive ALPPS stage I surgery, and receive ALPPS stage II surgery 3-6 weeks after stage I surgery.
  Interventions: Procedure: ALPPS surgery

INTERVENTIONS:
Drug: Tislelizumab — In experimental group, patients who meet the inclusion criteria will receive ALPPS stage I surgery, treated with Tislelizumab 2-4 weeks after stage I surgery, and receive ALPPS stage II surgery 2-4 weeks after Tislelizumab treatment, and treated with Tislelizumab q3W 6-12 months after stage II surgery.
  Arms: Alpps plus Tislelizumab group
Procedure: ALPPS surgery — In experimental group, patients who meet the inclusion criteria will receive ALPPS stage I surgery, and receive ALPPS stage II surgery 4-8 weeks after stage I surgery; In control group, patients who meet the inclusion criteria will receive ALPPS stage I surgery, and receive ALPPS stage II surgery 3-6 weeks after stage I surgery.

SUMMARY:
Study design: Prospective, single-center, phase IIa clinical trial; Primary endpoint: Recurrence free survival; Secondary endpoints: Safety, overall survival; Main characteristics of patients: Liver malignancy, required (extended) hemihepatectomy, insufficient liver reserve; Study approaches: The experimental group is treated with ALPPS combined with Tislelizumab, and the control group was treated with ALPPS; Sample size: 20 (10:10); Study process: In experimental group, patients who meet the inclusion criteria will receive ALPPS stage I surgery, treated with Tislelizumab 2-4 weeks after stage I surgery, and receive ALPPS stage II surgery 2-4 weeks after Tislelizumab treatment, and treated with Tislelizumab q3W 6-12 months after stage II surgery; In control group, patients who meet the inclusion criteria will receive ALPPS stage I surgery, and receive ALPPS stage II surgery 3-6 weeks after stage I surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤70 years;
2. ECOG physical condition score: 0~1;
3. Clinical/pathological diagnosis of primary liver cancer or intrahepatic metastatic colorectal cancer;
4. Clinical evaluation requires (extended) hemihepatectomy;
5. Liver function Child A level
6. sFLR < 30%
7. The main organs function well, and the examination indicators meet the following requirements:

   Routine blood tests:

   Hemoglobin ≥90 g/L (no blood transfusion within 14 days); Neutrophil count ≥1.5×10^9/L; Platelet count ≥80×10^9/L;

   Biochemical examination:

   Total bilirubin ≤2×ULN (upper normal value); ALT or AST ≤ 2.5×ULN; Endogenous creatinine clearance ≥ 50 mL /min (Cockcroft-Gault formula);
8. Sign the informed consent voluntarily;
9. Good compliance, and family members willing to cooperate with follow-up.

Exclusion Criteria:

1. Presence of extrahepatic organ/distant lymph node metastasis;
2. Hilar lymph node metastasis cannot be radically resected;
3. Patients with intrahepatic metastatic colorectal cancer had received second-line or above systemic therapy;
4. Other uncured malignant tumors;
5. Pregnant or lactating women who are pregnant during the study period need to withdraw from the clinical trial;
6. Concurrent use of any other antitumor therapy in patients with primary liver cancer;
7. Patients with intrahepatic metastatic colorectal cancer have been treated with antitumor therapy in addition to primary surgery and standard first-line/second-line therapy;
8. Patients with a known history of other systemic serious diseases before screening;
9. Long-term unhealed wounds or incomplete healing fractures;
10. Previous organ transplantation history;
11. Having a history of abuse of psychotropic substances and being unable to quit or having mental disorders;
12. A history of immune deficiency or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
13. Concomitant conditions that, in the investigator's judgment, seriously endanger the patient's safety or affect the patient's completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
recurrence free survival | 6 weeks
  recurrence free survival

SECONDARY OUTCOMES:
safety (incidence of adverse events and serious adverse events) | 3 weeks
  incidence of adverse events and serious adverse events
overall survival | 6 weeks
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China